CLINICAL TRIAL: NCT01765621
Title: Clinical and Economic Impact of a Web Based, Electronic Medical Record Interfaced Electronic Decision Support System Incorporating Pharmacogenetic Evaluation for Physicians Intended, Mainly for Drug-drug Interaction. A Controlled Study in an Ambulatory Health Maintenance Organization Population
Brief Title: Clinical and Economic Impact of an Electronic Medical Record Interfaced Decision Support System Reinforced With Patient Specific Pharmacogenetic Data for Minimizing Severe Drug-Drug Interactions
Acronym: DDI+
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leumit Health Services (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: LHS022013
Record Dates: First submitted 2013-01-09; First posted 2013-01-10 (Estimated); Last update posted 2014-10-21 (Estimated); Status verified 2014-10

CONDITIONS: Healthcare
Keywords: health care expenditure; drug drug interactions; electronic decision support systems; pharmacogenetics; Potential Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- DDI+ and Pharmacogenetic data (Experimental): DDI+ System and Pharmacogenetic data
  Interventions: Other: DDI+ System and Pharmacogenetic Data
- Standard Care (No Intervention): Control

INTERVENTIONS:
Other: DDI+ System and Pharmacogenetic Data
  Arms: DDI+ and Pharmacogenetic data

SUMMARY:
Leumit Health Services, an health maintenance organization operating in Israel, will incorporate a web-based, decision support system for handling drug-drug interactions and drug information, termed DDI+ reinforced with patient specific pharmacogenetic data. The investigators hypothesize that implementing such a system will reduce health-care expenditures (e.g., hospital admissions, referrals to ERs, Imaging procedures).

ELIGIBILITY:
Inclusion Criteria:

* Number of chronic concomitant drugs ≥5
* treated with 1 or more drugs with a well established interaction with 1 or more of the following CYP450 enzymes: 2c9, 2c19, 2d6

Exclusion Criteria:

* Patients diagnosed with HIV/AIDS, and/or viral hepatitis B or C

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 973 (Actual)
Dates: Start 2013-01; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Hospital Admissions | up to 12 month post initiation

CONTACTS AND LOCATIONS:
Locations (1):
- Leumit Health Services, Tel Aviv, Israel